CLINICAL TRIAL: NCT04679883
Title: A Phase 2 Multicenter, Randomized, Double-blinded, Placebo-controlled Trial to Evaluate the Efficacy and Safety of GLH8NDE in Patients With Dry Eye Disease
Brief Title: Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of GLH8NDE in Patients With Dry Eye Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLH8NDE-201
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GLH8NDE 5% and GLH8NDE Placebo (Experimental): Three times each 1 drop a day, total 6 times 1 drop of GLH8NDE 5% and GLH8NDE Placebo
  Interventions: Drug: 5% GLH8NDE; Drug: Placebo
- GLH8NDE 5% (Experimental): Total 6 times 1 drop of GLH8NDE 5%
  Interventions: Drug: 5% GLH8NDE
- GLH8NDE Placebo (Placebo Comparator): Total 6 times 1 drop of GLH8NDE Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5% GLH8NDE — 5% GLH8NDE as eye drops
  Arms: GLH8NDE 5%; GLH8NDE 5% and GLH8NDE Placebo
Drug: Placebo — Placebo as eye drops
  Arms: GLH8NDE 5% and GLH8NDE Placebo; GLH8NDE Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled phase 2 clinical trial to evaluate the efficacy and safety of GLH8NDE in patients with Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject who is the age of older than 19 years at the screeing visit
* Subject who has symptom at least one or more as below for six months(Irritation, foreign body sensation, burning, mucus discharge, blurring, itching, photophobia, tired or heavy feeling and pain)
* Subject with dry eye syndrome who meet all of the following criteria among the left and/or right eyes at the time of screening and baseline visit.

  1. Over six grade as fluorescein corneal staining by National Eye Institute scale
  2. Schirmer I test ≤ 10 mm/5 min.
  3. TFBUT ≤ 6 seconds
* At the screening and baseline visit, the intraocular pressure(IOP) of both eyes is more than 5 mmHg and below 22 mmHg
* At the screening and baseline visit, biocular best corrected visual acuity(BCVA) are over 0.2(=+0.7 logMAR or Snellen 20/100)
* At the baseline visit, over 80% administration compliance during run-in period as placebo in single blind
* Subject who signed and dated the informed consent form after understanding fully to hear a detailed explanation in the clinical trial

Exclusion Criteria:

* Ophthalmic diseases that may confuse the interpretation of clinical trial results, such as clinically significant corneal surface disease, abnormal corneal sensitivity, and abnormal tearing
* Subject with wounds caused by refractive surgery such as LASIK surgery (However, if it does not affect the clinical trial compliance and result evaluation according to the investigator's judgment, participation is possible.)
* Subject with the following concomitant diseses at screening visit.

  1. Eyelid disease (blepharopathy, blepharolysis, valgus, varus valgus, etc.), conjunctival relaxation, cataracts, and eye diseases requiring treatment
  2. Sjogren's syndrome and secondary Sjogren's syndrome (rheumatoid arthritis, systemic lupus erythematosus, etc.)
  3. Diabetes not controlled despite appropriate treatment (hemoglobin A1c (HbA1c)> 9%)
  4. Subject with the following systemic diseases that are not controlled High blood pressure that is not controlled despite administration of antihypertensive drugs (systolic blood pressure (SBP)/diastolic blood pressure (DBP)>160/100 mmHg) Clinically significant cardiopulmonary disease despite appropriate treatment
  5. Acute active hepatitis A, active hepatitis B or C
* Subject with the following medical history (including surgical history) at screening visit

  1. Organ transplant or bone marrow transplant
  2. History of known immunodeficiency disease or human immunodeficiency virus (HIV) infection
  3. Ophthalmic surgery within 1 year before screening (including LASIK/LASEK surgery)
  4. Subject who has undergone punctal occlusion and have not passed 12 weeks from the time point below.

After punctal cauterization using electrocautery. After inserting a permanent, semi-permanent punctal plug. If a temporary punctal plug is inserted, remove the punctal plug.

* Subject who has administered the following drugs before the clinical trial or who need to be administered during the clinical trial.

  1. Cyclosporine eye drops within 6 weeks before screening
  2. Ophthalmic solutions or antibiotics due to blepharitis, meibomian gland disease, herpes zoster, and eye infection within 6 weeks before screening
  3. Drugs that cause dry eye within 6 weeks before screening (anticholinergics, isotretinoin, etc.)
  4. Oral aspirin or drugs containing aspirin within 6 weeks before screening
  5. Contains corticosteroids, mast cell stabilizers, antihistamines, anti-inflammatory drugs (NSAIDs, etc.), gamma linolenic acid, or omega-3 fatty acids within 6 weeks before screening
  6. Other ophthalmic solutions within 3 days before screening
* Subject who wears contact lenses within 1 week before screening or who needs to wear them during the clinical trial
* Subject with alcoholism or drug abuse history within 1 year before screening
* Pregnant women, lactating women, and those who disagree with appropriate contraception during the clinical trial (visit 1 to visit 6)
* Subject with hypersensitivity to investigator's drugs or their excipients
* Subject who participated in other clinical trials within 4 weeks before screening and received/received investigator's drug or clinical trial medical devices
* Subject judged by other investigators to be inappropriate to participate in this clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
The change of Total Corneal Staining Score (TCSS) | Between 1 day before first IP administration and 4 weeks
  To 4 weeks after baseline visit using NEI scale (total between 0 and 15 scores)

SECONDARY OUTCOMES:
The change of Total Corneal Staining Score (TCSS) | Between 1 day before first IP administration and 2, 8, 12 weeks
  To 2, 8, 12 weeks after baseline visit using NEI scale (total between 0 and 15 scores, higher scores mean a worse outcome)
The change of Inferior Corneal Staining Score (ICSS) | Between 1 day before first IP administration and 2, 4, 8, 12 weeks
  To 2, 4, 8, 12 weeks after baseline visit using NEI scale (total between 0 and 15 scores, higher scores mean a worse outcome)
The change of Conjunctival Staining Score | Between 1 day before first IP administration and 2, 4, 8, 12 weeks
  To 2, 4, 8, 12 weeks after baseline visit using NEI scale (total between 0 and 18 scores, higher scores mean a worse outcome)
The change of Tear Film Break-up time(TFBUT) | Between 1 day before first IP administration and 2, 4, 8, 12 weeks
  To 2, 4, 8, 12 weeks after baseline visit
The change of Schirmer I test | Between 1 day before first IP administration and 2, 4, 8, 12 weeks
  To 2, 4, 8, 12 weeks after baseline visit
The change of 5-item dry questionnaire (DEQ-5) | Between 1 day before first IP administration and 2, 4, 8, 12 weeks
  To 2, 4, 8, 12 weeks after baseline visit (total between 0 and 22 socres, higher scores mean a worse outcome)
The change of Ehlers-Danlos Syndrome (EDS) by Visual Analogue Scale (VAS) | Between 1 day before first IP administration and 2, 4, 8, 12 weeks
  To 2, 4, 8, 12 weeks after baseline visit (total between 0 and 100 scores, highter scores mean a worse outcome)
The change of Ccular Discomfort Score(ODS) | Between 1 day before first IP administration and 2, 4, 8, 12 weeks
  To 2, 4, 8, 12 weeks after baseline visit (total 0 and 4 scores, higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea